CLINICAL TRIAL: NCT02678013
Title: Radiofrequency Ablation Combined With Highly-purified CTL vs. Radiofrequency Ablation Alone for Recurrent HCC
Brief Title: RFA+Highly-purified CTL vs. RFA Alone for Recurrent HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ming Kuang (Other)
Responsible Party: Sponsor-Investigator, Ming Kuang, Ph.D.,M.D., Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 004
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiofrequency ablation(RFA) (Experimental): RFA was performed according to the Guidelines of Radiofrequency Ablation Therapy for Liver Cancer: Chinese Expert Consensus Statement issued by the Chinese Society of Liver Cancer and Chinese Society of Clinical Oncology RFA was performed under real-time ultrasound guidance. RFA was performed by using a commercially available Cool-tipTM RFA system (Valleylab, Boulder, CO, USA), or a RF 2000 system (Radio-Therapeutics Mountain View, CA). Grounding was achieved by attaching 2 pads to the patient's back or legs.
  Interventions: Procedure: RFA
- RFA+CTL (Active Comparator): RFA was performed the same as RFA Arm.Peripheral blood (20-30mL) for manufacturing the individualized highly-purified CTL agent was collected from the respective patients who were randomized to the immunotherapy group before starting treatment. The highly-purified CTL agent was prepared at a central manufacturing facility. Patients in the immunotherapy group received 5*10E9 of the highly-purified CTL agent intravenously over 60 minutes without any premedication and then were observed for at least 30 minutes. They were scheduled to receive highly-purified CTL: 4-6 treatments at a frequency of once two-week during 6 months after receiving RFA, followed by 6-9 treatments during 6 months to 2 years after receiving RFA.
  Interventions: Procedure: RFA+highly-purified CTL

INTERVENTIONS:
Procedure: RFA — Radiofrequency ablation(RFA)for small recurrent HCC
  Arms: Radiofrequency ablation(RFA)
Procedure: RFA+highly-purified CTL — Radiofrequency ablation(RFA) plus highly-purified CTL for small recurrent HCC
  Arms: RFA+CTL

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common and the third leading cause of cancer-related death worldwide. Recurrence of tumor within the liver remnant is common, with a reported 5-year recurrence rate of 70%. Repeat hepatectomy is an effective treatment for intrahepatic HCC but with a small proportion of resection rate because of the poor functional liver reserve and postoperative complications. Radiofrequency ablation(RFA) is becoming the main effective treatment for small HCC (≤5.0cm). The efficacy of RFA for recurrent HCC has been reported to be comparable to those achieved by surgery with minimal, but higher local recurrence rate after RFA. It has been reported that immunotherapy in patients who underwent curative treatment for HCC, adjuvant immunotherapy with activated CIK cells increased recurrence-free and overall survival. But there is little evidence for adjuvant immunotherapy of recurrence HCC. Cytotoxic T lymphocytes(CTL), a kind of effective T cells that specific recognizing and killing antigen targeted cells through cloning amplification after receiving antigen information from antigen presented cell and playing key role to clear cancerous cells. So our hypothesis is that RFA combined with immunotherapy (Highly-purified CTL) is superior to RFA for recurrent HCC. The aim of this prospective study is to compare the outcome of RFA combined with immunotherapy (Highly-purified CTL) with RFA for small recurrent HCC after partial hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years;
2. recurrence of HCC 12 months after initial hepatectomy;
3. no other treatment received except for the initial hepatectomy;
4. single tumor≤5.0cm in diameter; or 2-3 lesions each≤3.0cm;
5. lesions visible on ultrasound and with an acceptable and safe path between the lesion and the skin as shown on ultrasound;
6. no severe coagulation disorders (prothrombin activity<40% or a platelet count<40,000/mm3);
7. Eastern Co-operative Oncology Group performance(ECOG) status 0-1.

Exclusion Criteria:

1. Pregnant women, breastfeeding women or plan pregnancy for the future 2 years;
2. The presence of vascular invasion or extrahepatic spread onimaging;
3. Usage of strong immunosuppressive agents such as corticosteroids, cyclosporine A within six months or longer;
4. HIV antibody or HCV antibody positive;
5. Immunodeficiency diseases or autoimmune diseases (such as rheumatoid arthritis, Buerger's disease, multiple sclerosis and type 1 diabetes);
6. Suffering with cancers (except skin cancer, prostate cancer or cervical carcinoma in situ) at the enrolling time or 5 years before;
7. Suffering with other organ failure;
8. Suffering with severe mental illness;
9. Drug addiction (including alcohol) for 1 year before the enrolling time;
10. Participate in other Clinical trials within three months prior to 3 months before the enrolling time;
11. Other researchers believe that the patient is not fit for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2016-02; Primary Completion 2020-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 2 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, Ph.D., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Zhen-Wei Peng, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Background] Lee JH, Lee Y, Lee M, Heo MK, Song JS, Kim KH, Lee H, Yi NJ, Lee KW, Suh KS, Bae YS, Kim YJ. A phase I/IIa study of adjuvant immunotherapy with tumour antigen-pulsed dendritic cells in patients with hepatocellular carcinoma. Br J Cancer. 2015 Dec 22;113(12):1666-76. doi: 10.1038/bjc.2015.430. Epub 2015 Dec 10. PMID 26657650
- [Background] Harding JJ, El Dika I, Abou-Alfa GK. Immunotherapy in hepatocellular carcinoma: Primed to make a difference? Cancer. 2016 Feb 1;122(3):367-77. doi: 10.1002/cncr.29769. Epub 2015 Nov 5. PMID 26540029